CLINICAL TRIAL: NCT05075785
Title: National Epidemiological Cohort to Evaluate Covid-19 Respiratory Sequelae: a French Pneumologist Collaboration.
Brief Title: Covid-19 Respiratory Sequelae French Cohort
Acronym: PNEUMOCOVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Cabinet Medical valenciennes (Unknown); CH Aix (Unknown); hopital privé de bois bernard (Unknown); Clinique La Croix du Sud (Unknown); University Hospital, Bordeaux (Other); Hopital Forcilles (Other); Hopital d'instructions des armées (Unknown); Hôpital Européen Marseille (Other); Rennes University Hospital (Other); Clinique Saint Augustin (Unknown); Delafontaine Hospital (Other); Centre Hospitalier Universitaire de Saint Etienne (Other); Centre Hospitalier de Troyes (Other); Centre Hospitalier le Mans (Other); University Hospital, Clermont-Ferrand (Other); University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0135
Record Dates: First submitted 2021-10-12; First posted 2021-10-13 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: COVID-19; Fibrosis; Cohort; Follow-up; Sequelae; Spirometry DLCO
Keywords: COVID-19; Fibrosis; cohort; follow-up; Sequelae; spirometry DLCO
MeSH Terms: conditions — COVID-19; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As the investigators need data on long term outcome of Covid-19, especially respiratory sequelae, a national cohort is required. To better evaluate the potential respiratory sequelae after SARS-CoV-2 infection, it is fundamental to include patients with different management at the acute phase of the Covid-19: ambulatory management, hospitalization in non ICU and in ICU units. That is why the investigators will conduct a national cohort study with all components of french pneumology which will give the investigators the opportunity to include patients in general hospital, in university hospital and in private structure. As it is a "real life" study, the investigators will include all patients who will have a consultation with a pneumologist for an evaluation 5 to 7 months after a Covid-19 infection whatever their acute disease management. The investigators will collect all available data on Covid-19 acute phase, on patients characteristics and comorbidities, on persistent symptoms after Covid-19, on exams results during the outcome evaluation (CT-scan, 6 min walk test, spirometry and DLCO, blood gas, VO2 max if realized).

ELIGIBILITY:
Inclusion Criteria:

* adults, older than 18
* SARS-CoV-2 infection confirmed by polymerase chain reaction (PCR) in nasopharyngeal swab in patients who are evaluated by a pneumologist 5 to 7 months after their Covid-19 disease

Exclusion Criteria:

* patients for whom follow-up would be difficult owing to psychotic disorder
* dementia
* patients who have declined to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As it is a "real life" study, the investigators will include all patients who will have a consultation with a pneumologist for an evaluation 5 to 7 months after a Covid-19 infection whatever their acute disease management.
  This is a cohort study with collection of different data. The proposed follow-up of these patients is the recommended follow-up of the french respiratory society. But, as it is a real life study, no exams are mandatory.
Sampling Method: Non-Probability Sample
Enrollment: 2933 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Variation of vital capacity at 5 months after Covid-19 episode | at 5 months
Variation of vital capacity at 7 months after Covid-19 episode | at 7 months
DLCO alteration at 5 months after Covid-19 episode | at 5 months
DLCO alteration at 7 months after Covid-19 episode | at 7 months
desaturation during the "6 min walk test" | at 5 months
desaturation during the "6 min walk test" | at 7 months

SECONDARY OUTCOMES:
Variation of FEV1 spirometry parameters | at 5 months
Variation of FEV1 spirometry parameters | at 7 months
Variation of VC spirometry parameters | at 5 months
Variation of VC spirometry parameters | at 7 months
Variation of FVC spirometry parameters | at 5 months
Variation of FVC spirometry parameters | at 7 months
Variation of DLCO spirometry parameters | at 5 months
Variation of DLCO spirometry parameters | at 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No